CLINICAL TRIAL: NCT04864600
Title: CANDLE - A Study of Acute Health Effects of Exposure to Particles Generated by Candles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Lund University (Other); University of Copenhagen (Other); Danish Technological Institute (Unknown); ASP-HOLMBLAD A/S (Unknown); COOP Denmark (Unknown); Danwax (Unknown); Liljeholmens Stearinfabrik (Unknown); Promol (Unknown); European Candle Association (Unknown)
Responsible Party: Principal Investigator, Torben Sigsgaard, Professor and medical doctor, University of Aarhus
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 201100
Record Dates: First submitted 2020-11-04; First posted 2021-04-29 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Inflammatory Response; Symptoms and Signs
Keywords: Stearin candle; Health effects; Inflammation; Asthmatics; Particle contamination; Indoor air; Pollutant
MeSH Terms: conditions — Signs and Symptoms; Inflammation; Asthma

STUDY DESIGN:
Intervention Model Description: A randomized cross-over double-blind study under controlled conditions in a climate chamber having three different exposures; A) a standard (Scandinavian) stearin candle, B) a modified low emitting version of the same candle, and C) clean air
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Stearin Candle (Active Comparator): Several candles will be lit. We will be using realistic burning cycles i.e. burning candles which extinguish and new ones being lit.
  Interventions: Other: Candle 1
- Modified low emission candle (Experimental): Several candles will be lit. We will be using realistic burning cycles i.e. burning candles which extinguish and new ones being lit.
  Interventions: Other: Candle C
- Clean Air (No Intervention): No candles in the chamber.

INTERVENTIONS:
Other: Candle C — Burning candles will produce particulate air pollution being passed on an exposure chamber where the participants will be sitting for 5 hours.
  Arms: Modified low emission candle
Other: Candle 1 — Burning candles will produce particulate air pollution being passed on an exposure chamber where the participants will be sitting for 5 hours.
  Arms: Standard Stearin Candle

SUMMARY:
INTRODUCTION: Particle contamination is suggested to have substantial negative effects on health, with candles emitting huge amount of particles, thus being one of the largest contributors to indoor air pollution. Chronic low levels of exposure to indoor particles over time is an important risk factor for the health of the population as a whole and it becomes particularly important for vulnerable groups like people suffering from respiratory diseases such as asthma.

AIM: In a randomized controlled cross-over trial the difference in health effects between two candles I) a standard candle and II) a low emission candle modified from the standard candle is studied.

DETAILED DESCRIPTION:
INTRODUCTION; Particle contamination is suggested to have substantial negative effects on health, with candles emitting the huge amount of particles, thus being one of the largest contributors to indoor air pollution. Chronic low levels of exposure to indoor particles over time is an important risk factor for the health of the population as a whole and it becomes particularly important for vulnerable groups like children and the elderly or people already suffering from allergies and respiratory diseases such as asthma.

AIM: To study the difference in health effects between two candles I) a standard candle and II) a low emission candle modified from the standard candle. The following hypothesis will be examined: Short-term exposure to particles generated by the standard candle is associated with more objectively measurable effects in metabolomics inflammation compared to exposure to modified low-emission candle particles.

METHODS: Separated by two weeks 20 young asthmatics will be exposed in a randomized cross-over double-blind study under controlled conditions in a climate chamber to three different exposures; A) a standard (Scandinavian) stearin candle, B) a modified low emitting version of the same candle, and C) clean air from the adjacent chamber. The experiment will be carried out in groups of 3-6 participants.

MEASUREMENTS: TSI P-TRAK Ultrafine Particle Counter and SMPS will be used for particle counts. Health effects, including spirometry and fraction of exhaled nitric oxide (FeNO) will be evaluated in relation to local and systemic effects prior to, right after and 24 h. after exposure.

ANALYSIS: Mixed methods approach taking both time and exposure into account.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-25
* Medically treated / physician diagnosed mild seasonal asthma GINA guidelines step 1 or 2 (https://ginasthma.org/)
* Never smoker or ex-smoker ≥ 6 months
* Allergy > 1 common allergy

Exclusion Criteria:

* Any other disease that could influence the study parameters
* Conditions that prevent safe access to the climate chambers (such as claustrophobia)
* Perennial asthma
* Need for continuous medical treatment for asthma
* Pregnancy

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Particles in Exhaled Air (Surfactant Protein A & Albumin) | At baseline (0 hour), after exposure (5 hours), and the day after exposure (24 hours)
  PExA: Subjects performed repeated breath maneuvers allowing for airway closure and re-opening, and exhaled particles were optically counted and collected on a membrane using the PExA® instrument set-up

SECONDARY OUTCOMES:
Change in Lung Function (FEV1 & FVC) | At baseline (0 hour), after exposure (5 hours), and the day after exposure (24 hours)
  Spirometry
Change in Fractional exhaled nitric oxide (FENO) | At baseline (0 hour), after exposure (5 hours), and the day after exposure (24 hours)
  NIOX VERO system; Aerocrine AB, Sweden
Change in white blood cells in Blood | At baseline (0 hour), after exposure (5 hours), and the day after exposure (24 hours)
  White blood cells
Change in Endothelial Progenitor Cells (EPCs) in Blood | At baseline (0 hour), after exposure (5 hours), and the day after exposure (24 hours)
  Endothelial progenitor cells (EPC) further divided into early and late EPCs
Change in inflammatory markers in Blood | At baseline (0 hour), after exposure (5 hours), and the day after exposure (24 hours)
  Interleukin 8, interleukin 1
Change in biomarkers in Blood | At baseline (0 hour), after exposure (5 hours), and the day after exposure (24 hours)
  Metabolomics
Change in nasal volume (using Acoustic rhinometry) | At baseline (0 hour), after exposure (5 hours), and the day after exposure (24 hours)
  Acoustic rhinometry is used to assess the nasal cross sectional area and volume. The left and right nasal cavity were studied alternatively until three reproducible measurements were obtained. The minimum cross sectional cavity area is calculated from the means of the measurements. By integration of the area-distance curve, the sum of the volume 2 to 4 (vol2-4) from the nostril is determined on both sides.
Change in biomarkers in Saliva Sample | after exposure (5 hours), and the day after exposure (24 hours)
  An oral svap from Salivette was placed in the mouth of the participant to collect saliva by gently chewing the swab for one minute. Afterwards the saturated swab was removed to the suspended insert and closed firmly with a lid. Then the sample was transferred to a freezer and stored for -80 C until further analysis. The sample will be analyzed for biomarkers (amylase, cortisol, substance P, lysozyme and secretory IgA. (same unit measure))
ReCIVA | At baseline (0 hour), after exposure (5 hours), and the day after exposure (24 hours)
  Sampling of VOCs and particles in exhaled air. Breathing through a mask for 10-15 minutes makes it possible to collect VOCs and particles into tenax air sampling tubes.
Change in Subjective Symptoms | Every 30 minute during 5 hours of exposure
  n the exposure chamber participants are asked to fill out a symptom questionnaire every 30 minute regarding their well-being and experienced symptoms in eyes, nose and throat. The participants are asked to score their evaluation / rate the strength of symptoms on a Linear Numeric Scale from 0-10, with 10 being worst. Health effects are evaluated in relation to rated changes in symptoms
Heart rate using a Fitbit | From exposure start until the morning after exposure (in total 24 hours)
  Using a Fitbit watch participants' heart rate is measured.
Sleep quality using a Fitbit | during 48 hours
  Using a Fitbit watch participants' sleep quality is measured.

CONTACTS AND LOCATIONS:
Overall Officials: Torben Sigsgaard, Prof., Principal Investigator — University of Aarhus
Locations (1):
- Climate Chambers, Dept. Public Health, Aarhus University, Aarhus, Central Region Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No